## Official Title:

Compensatory Kinematic Movements in Various Directions After Stroke

## **NCT Number:**

NCT05683158

## **Document Date:**

July 19, 2022

## **Statistical Analysis**

Statistical analyses were performed using various methods to comprehensively evaluate the data. For comparing demographic and clinical characteristics between the two groups, both chi-square test and t-test were employed.

The main analysis utilized two-way mixed-design analyses of variance, conducted independently for each variable. This analysis incorporated three levels as the within-subject factor and the participant group (healthy, stroke) as the between-subject factor. To account for multiple comparisons, Bonferroni post-hoc tests were performed. All statistical analyses were conducted using a significance level ( $\alpha$ ) of p < 0.05.

Sample size determination was carried out using G\*Power V.3.1 software (Franz Paul, Kiel, Germany) (Faul et al., 2007). The calculation parameters included an effect size (d) of 1.9, significance level ( $\alpha$ )  $\leq$  0.05, power = 0.8, and type II error ( $\beta$ ) = 0.2, following the methodology of previous research (Machado et al., 2019).